CLINICAL TRIAL: NCT00579891
Title: Tissue and Serum Collection From Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 89-006
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; tissue collection
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum tissue

SUMMARY:
To establish a serum and tissue bank with specimens form patients with colorectal cancer, for subsequent immunological and biochemical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be undergoing surgery for resection of their primary tumor, resection of hepatic metastases, or hepatic artery catheter and pump implant for unresectable hepatic metastases.
* For and tumor specimen removed at surgery ,the lesion must be large enough to allow for routine pathological analysis, with excision from residual otherwise discarded material for the tumor bank.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Colorectal cancer patients undergoing surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 726 (Actual)
Dates: Start 1989-03-28 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
establish a serum and tissue bank | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Philip Paty, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org